CLINICAL TRIAL: NCT05826834
Title: An Investigation of Ball Rolling Effects on Trigger Points
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Memorial University of Newfoundland (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Principal Investigator, Saman Anvar, Principal Investigator, Memorial University of Newfoundland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20211162
Record Dates: First submitted 2023-03-23; First posted 2023-04-24 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Trigger Point Pain, Myofascial
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ball rolling (Experimental): The ball-rolling group will be asked to roll the ball on the trapezius muscle.
  Interventions: Device: ball-rolling (Myostorm ball)
- Control (No Intervention): The control group with no intervention

INTERVENTIONS:
Device: ball-rolling (Myostorm ball) — the intervention group
  Arms: Ball rolling

SUMMARY:
The current study aims to examine the potential effects of rolling a Myostorm ball on the trigger points in the upper back muscles.

DETAILED DESCRIPTION:
The investigators will ask the participants to attend the laboratory in two sessions. They will seek the tender spots on the trapezius muscle. Then the participants will be asked to roll a Myostorm ball ( a small hard ball made of plastic with a layer of soft material cover) on their affected muscles. They will be tested for pain-pressure threshold (PPT), shoulder range of motion, electromyography (EMG), and force before and after the manipulation.

ELIGIBILITY:
Inclusion Criteria:

* trigger points on the trapezius muscle

Exclusion Criteria:

* back injury

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Range of Motion before ball rolling | 3 minutes before the intervention (Ball-rolling)
  the range of motion in the shoulder joint
Pain pressure threshold before ball rolling | 3 minutes before the intervention (Ball-rolling)
  the measurement of the pain pressure threshold on the trapezius muscle using Lafayette Muscle Tester; A hand-held algometer will be applied on the participant's skin and an incremental pressure will be applied until the participant notify the experimenter to stop. The pain pressure threshold will be reported in kilogram/cm2.
Range of Motion after ball rolling | up to 3 minutes after the intervention (Ball-rolling)
  the range of motion in the shoulder joint
Pain pressure threshold after ball rolling | up to 3 minutes after the intervention (Ball-rolling)
  the measurement of the pain pressure threshold on the trapezius muscle using Lafayette Muscle Tester; A hand-held algometer will be applied on the participant's skin and an incremental pressure will be applied until the participant notify the experimenter to stop. The pain pressure threshold will be reported in kilogram/cm2.

IPD SHARING:
Plan to Share IPD: Yes
The data will be kept confidential, and the participant codes will be used to link individual data across the experiment sessions. Data will be stored physically and digitally in Dr. Behm's office.
  Every reasonable effort will be made to ensure the participants' anonymity. They will not be identified in publications without their explicit permission. All data will be collected independently and kept confidential.
  All data will be stored in hardcopy and password-protected digital copy in Dr. David Behm's office at the Memorial University of Newfoundland. Consent forms will be stored separately from participant data in a locked cabinet in Dr. David Behm's office. Data access will be limited only to our research team members.
  Data potentially may be published in an online journal article. Published data will contain no personally identifying information.
Supporting Information: CSR
Time Frame: Data will be kept for at least five years, as Memorial University's policy on Integrity in Scholarly Research requires.